CLINICAL TRIAL: NCT04989803
Title: A Phase 1/2 Open-label, Multicenter Study Evaluating the Safety and Efficacy of KITE-363 or KITE-753, Autologous Anti-CD19/CD20 CAR T-cell Therapies, in Subjects With Relapsed and/or Refractory B-cell Lymphoma
Brief Title: Study of KITE-363 or KITE-753 in Participants With Relapsed and/or Refractory B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-499-0150; 2020-000562-41 (EudraCT Number); 2024-511616-24 (Other: CTIS Number)
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Relapsed and/or Refractory B-cell Lymphoma
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase 1 a/b: KITE-363 (Experimental): Phase 1a (Dose escalation): Participants with r/r large B-cell lymphoma will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single target starting dose of KITE-363 chimeric antigen receptor (CAR) transduced autologous T cells. Based on dose limiting toxicities (DLTs) observed in the first cohort, additional participants will be enrolled and administered escalating dose of KITE-363.
  Phase 1b (Dose expansion): After completion of dose escalation, additional participants with r/r B-cell lymphoma across different disease indications will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single dose of KITE-363 at 1 or more dose-level deemed to be tolerable.
  [Recruitment completed for this arm]
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: KITE-363
- Phase 1 a/b: KITE-753 (Experimental): Phase 1a (Dose escalation): Participants with r/r large B-cell lymphoma will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single target starting dose of KITE-753 chimeric antigen receptor (CAR) transduced autologous T cells. Based on dose limiting toxicities (DLTs) observed in the first cohort, additional participants will be enrolled and administered escalating dose of KITE-753.
  Phase 1b (Dose expansion): After completion of dose escalation, additional participants with r/r B-cell lymphoma across different disease indications will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single dose of KITE-753 at 1 or more dose-level deemed to be tolerable.
  [Recruitment open for frontline LBCL and r/r MCL for this arm]
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: KITE-753
- Phase 2: KITE-753 (Experimental): Participants with r/r large B-cell lymphoma who have received at least 2 prior lines of systemic therapy will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single target starting dose of KITE-753 chimeric antigen receptor (CAR) transduced autologous T cells /kg intravenously (IV).
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: KITE-753

INTERVENTIONS:
Drug: Cyclophosphamide — Lymphodepleting chemotherapy administered intravenously
Drug: Fludarabine — Lymphodepleting chemotherapy administered intravenously
Biological: KITE-363 — A single infusion of CAR-transduced autologous T cells administered intravenously
  Arms: Phase 1 a/b: KITE-363
Biological: KITE-753 — A single infusion of CAR-transduced autologous T cells administered intravenously
  Arms: Phase 1 a/b: KITE-753; Phase 2: KITE-753

SUMMARY:
The goal of this clinical study is to learn more about the safety and effectiveness of the study drugs, KITE-363 and KITE-753, in participants with relapsed and/or refractory B-cell lymphoma.

DETAILED DESCRIPTION:
Eligible study participants who have received IP administration with either KITE-363 or KITE-753 will transition to a separate Long-term Follow-up study (Study KT-US-982-5968) to complete the remainder of the 15-year follow-up assessments.

ELIGIBILITY:
Key Inclusion Criteria: for Phase 1a/b and Phase 2

* Relapsed and/or refractory B-cell lymphoma (R/R BCL).
* At least 1 measurable lesion.
* Adequate organ and bone marrow (BM) function.

Key Exclusion Criteria: for Phase 1a/b and Phase 2

- History of chimeric antigen receptor (CAR) therapy or other genetically modified T cell therapy.

* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (eg, cervix, bladder, or breast) unless disease free and without anticancer therapy (with the exception of hormonal therapy in the case of breast cancer) for at least 3 years.
* History of Richter's transformation of chronic leukemic lymphoma, small lymphocytic lymphoma, or lymphoplasmacytic lymphoma.
* History of allogeneic stem cell transplant (allo-SCT).
* Auto-SCT within 6 weeks before the planned KITE-363 or KITE-753 infusion.
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requires intravenous (IV) antimicrobials for management.
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B virus (HBV) hepatitis B surface (HBs) antigen (HBsAg) positive infection, or hepatitis C (anti-hepatitis C virus [HCV] positive) infection.
* Individuals with detectable cerebrospinal fluid (CSF) malignant cells or brain metastases or a history of central nervous system (CNS) lymphoma, primary CNS lymphoma, or spinal epidural involvement.
* History or presence of a CNS disorder.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, active arrhythmia, New York Heart Association Class II or greater congestive heart failure or other clinically significant cardiac disease within the 6 months before enrollment.
* Primary immunodeficiency.
* History of autoimmune disease resulting in or requiring systemic immunosuppression and/or systemic disease-modifying agents within the last 2 years.
* History of non-line associated, clinically significant deep-vein thrombosis or pulmonary embolism requiring therapeutic anticoagulation within the 6 months before enrollment.
* Females of childbearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Females who have undergone surgical sterilization or have been postmenopausal for at least 2 years are not considered to be of childbearing potential.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Percentage of Participants Experiencing Adverse Events Defined as Dose-limiting Toxicities (DLTs) After the Infusion of KITE-363 or KITE-753 | Up to 28 days
  DLTs are defined as the KITE-363-related or KITE-753-related events with onset within the first 28 days after the infusion of KITE-363 or KITE-753 respectively.
Phase 1b: Objective Response Rate (ORR) for KITE-363 and KITE-753 as per investigator's assessment. | Up to 15 years
  ORR is defined as the percentage of participants with a complete response (CR) or a partial response (PR) by the International Working Group (IWG) Lugano Response Criteria for Malignant Lymphoma (Cheson 2014) as determined by investigator assessment.
Phase 2: ORR as per central assessment for KITE-753 | Up to 15 years

SECONDARY OUTCOMES:
Phase 1a/b: Percentage of Participants Experiencing Adverse Events (AEs) After the Infusion of KITE-363 and KITE-753 | Up to 15 years
Phase 1a/b: Percentage of Participants Experiencing Serious AEs (SAEs) After the Infusion of KITE-363 and KITE-753 | Up to 15 years
Phase 1a/b: Time To Next Treatment (TTNT) for KITE-363 and KITE-753 | Up to 15 years
  TTNT is defined as the time from KITE-363 or KITE-753 infusion to the next anticancer treatment (including stem cell transplantation [SCT]) or death from any cause, whichever occurs first.
Phase 1a/b: Complete Response (CR) Rate for KITE-363 and KITE-753 | Up to 15 years
  CR rate is defined as the incidence of a CR by the IWG Lugano Response Criteria for Malignant Lymphoma (Cheson 2014) as determined by investigator assessment.
Phase 1a/b: Duration of Response (DOR) for KITE-363 and KITE-753 | Up to 15 years
  DOR is defined only for participants who experience an objective response and is the time from the first objective response to disease progression per the IWG Lugano Classification or death due to any cause, whichever occurs first.
Phase 1a/b: Progression-Free Survival (PFS) for KITE-363 and KITE-753 | Up to 15 years
  PFS is defined as the time of KITE-363 or KITE-753 infusion to disease progression per IWG Lugano Response Criteria for Malignant Lymphoma (Cheson 2014) or death from any cause, whichever occurs first.
Phase 1a/b: Overall Survival (OS) for KITE-363 and KITE-753 | Up to 15 years
  OS is defined as the time from KITE-363 or KITE-753 infusion to death from any cause.
Phase 1a/b: Percentage of Participants who Develop Antibodies to KITE-363 and KITE-753 Chimeric Antigen Receptor (CAR) T Cells | Enrollment; up to 12 months
Phase 1a/b: Levels of KITE-363 and KITE-753 CAR T Cells | Up to 15 years
Phase 1a/b: Peak Serum Levels of Key Analytes Homeostatic/Proliferative Cytokines: Interleukin (IL)-2, IL-7, and IL-15 | Up to 3 months
Phase 1a/b: Peak Serum Levels of Key Analytes Inflammatory/Immune Modulating Cytokines: IFN-γ, IL-6, IL-10, IL-17, IL-1RA, Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF), and Tumor Necrosis Factor-Alpha (TNF-α) | Up to 3 months
  IFN-γ=Interferon-Gamma, IL-1 Receptor Antagonist=IL-1RA
Phase 1a/b: Peak Serum Levels of Key Analytes Correlates of Acute Phase Response: C-Reactive Protein (CRP) | Up to 3 months
Phase 1a/b: Peak Serum Levels of Key Analytes Correlates of Acute Phase Response: Ferritin | Up to 3 months
Phase 1a/b: Peak Serum Levels of Key Analytes Correlates of Acute Phase Response: Soluble IL-2 Receptor Alpha (Sil-2Rα) | Up to 3 months
Phase 1a/b: Peak Serum Levels of Key Analytes Chemokines: IL-8, C-X-C Motif Chemokine Ligand-10 (CXCL-10), and Monocyte Chemotactic Protein-1 (MCP-1) | Up to 3 months
Phase 1a/b: Peak Serum Levels of Key Analytes Immune-Effector Molecules: Perforin, Granzyme A, and Granzyme B | Up to 3 months
Phase 2: CR rate for KITE-753 | Up to 15 years
Phase 2: DOR for KITE-753 | Up to 15 years
Phase 2: PFS for KITE-753 | Up to 15 years
Phase 2: OS for KITE-753 | Up to 15 years
Phase 2: Percentage of Participants Experiencing Adverse Events (AEs) After the Infusion of KITE-753 | Up to 15 years
Phase 2: Percentage of Participants Experiencing Serious AEs (SAEs) After the Infusion of KITE-753 | Up to 15 years
Phase 2: ctDNA MRD-Negative CR Rate of KITE-753 | Up to 15 years
Phase 2: Overall ctDNA MRD Negativity of KITE-753 | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (14):
- United States (10):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Stanford Cancer Institute, Stanford, California
  - Northside Hospital, Atlanta, Georgia
  - University of MD, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Wexner Medical Center - James Cancer Hospital, Columbus, Ohio
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Royal North Shore Hospital, St Leonards, New South Wales, Australia
- Universitatsklinikum Wurzburg, Würzburg, Germany
- Academisch Medisch Centrum, Amsterdam, Netherlands
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-499-0150